CLINICAL TRIAL: NCT04282174
Title: A Phase II Trial of CD34+ Enriched Transplants From HLA-Compatible Related or Unrelated Donors for Treatment of Patients With Hematologic Malignancies
Brief Title: CD34+ Enriched Transplants From HLA-Compatible Patients With Hematologic Malignancies
Acronym: 2019-KOE-001
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was split into two new studies before the first participant was enrolled.
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KOE-001
Record Dates: First submitted 2020-02-17; First posted 2020-02-24 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Hematologic Diseases; Hematologic Malignancy; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Myelogenous Leukemia; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Hematologic Diseases; Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bone Marrow Transplantation; Thiotepa; Cyclophosphamide; Busulfan; Melphalan; fludarabine

STUDY DESIGN:
Intervention Model Description: The two myeloablative conditioning regimens are:
  Regimen A: Hyperfractionated Total Body Irradiation/Thiotepa/Cyclophosphamide: 100 patients Regimen B: Busulfan/Melphalan/Fludarabine: 100 patients It is anticipated that the accrual will last five years. Patients will be followed for two years following transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Regimen A (Experimental): Regimen A: Hyperfractionated Total Body Irradiation/Thiotepa/Cyclophosphamide: Hyperfractionated total body irradiation to dose of 1375cGy fractions at 4-6 hour intervals three times a day for a total of 11 or 12 doses depending on age and disease risk, followed by Thiotepa 5mg/kg/day x 2 (or 10mg/kg/day x 1) and cyclophosphamide 60mg/kg/day x 2 (or Fludarabine 25mg/m2 x 5 if cyclophosphamide is contraindicated)
  Interventions: Device: CliniMACS; Procedure: Bone Marrow Transplant; Drug: Hyperfractionated Total Body Irradiation; Drug: Thiotepa; Drug: Cyclophosphamide
- Regimen B (Experimental): Regimen B: Busulfan/Melphalan/Fludarabine: Busulfan 0.8mg/kg/dose every six hours x 10-12 doses (depending on disease), Melphalan 70mg/m2/day x 2 and Fludarabine 25mg/m2/day x 5.
  Interventions: Device: CliniMACS; Procedure: Bone Marrow Transplant; Drug: Busulfan; Drug: Melphalan; Drug: Fludarabine

INTERVENTIONS:
Device: CliniMACS — allogeneic Human leukocyte antigen-compatible related or unrelated transplants of GCSF-mobilized peripheral blood stem cells depleted of T-cells by positive selection of CD34+ progenitor cells using the CliniMACS system
Procedure: Bone Marrow Transplant — Bone Marrow Transplant will come from either an HLA matched related sibling or HLA un-related donor
Drug: Hyperfractionated Total Body Irradiation — Hyperfractionated Total Body Irradiation is administered at a dose rate of < 20 cGy/minute. Doses of 125 cGy/fraction are administered at a minimum interval of 4 hours between fractions, three times/day for a total of 11 or 12 doses (1375 or 1500 cGy) over 4 days (Day -9, -8, -7 and -6).
  Arms: Regimen A
Drug: Thiotepa — Thiotepa: 5mg/kg/day IV over approximately 4 hr. daily x 2 (Day -5 and Day -4). If scheduling of transplant harvests requires, the dose of Thiotepa may be administered as a single dose of 10mg/kg/day x 1.
  Arms: Regimen A
Drug: Cyclophosphamide — Cyclophosphamide: 60 mg/kg/day I V over approximately 30 min daily x 2 days (d -3 and -2). Cyclophosphamide dosing will be adjusted if patient is > 125% of ideal body w eight and will be calculated based on adjusted ideal body weight, as per MCI standard of care guidelines.
  Arms: Regimen A
Drug: Busulfan — 0.8 mg/kg every 6 hours x 10 or 12 doses), (depending on disease) with dose modified
  Arms: Regimen B
Drug: Melphalan — Melphalan 70mg/m2/day x 2 days IV over 30 minutes. Dose should be adjusted if patient is > 125% ideal body weight and should be calculated on adjusted ideal body weight per MCI standard of care guidelines. Melphalan will be administered on Days - 7 and -6 for multiple myeloma patients.
  Arms: Regimen B
Drug: Fludarabine — Fludarabine 25mg/m2/days x 5 days IV over 30 minutes. Fludarabine may be adjusted in the case of renal toxicity.
  In select cases in which the peripheral blood stem cells must be harvested a day later than requested due to a scheduling issue with the donor or Stem Cell Processing Laboratory.
  Arms: Regimen B

SUMMARY:
This is a Phase II trial testing disease-specific myeloablative conditioning regimens for preparatory cytoreduction of patients receiving allogeneic HLA-compatible related or unrelated transplants of GCSF-mobilized peripheral blood stem cells (PBSC) depleted of T-cells by positive selection of CD34+ progenitor cells using the CliniMACS system. The CliniMACS Fractionation system is a method that positively selects CD34+ progenitor cells from PBSC by immunoadsorption of cells binding on anti CD34 monoclonal antibody to paramagnetic beads, which can then be isolated by passage through a magnetized column and released by agitation of beads. Two conditioning regimens have been used successfully with an alternative similar system, isolex, which is no longer being manufactured.

DETAILED DESCRIPTION:
For this trial, patients will be put into one of two myeloablative conditioning regimens, based on their disease, stage of disease, and dose of radiation accumulated in the course of treatment. Approximately twenty-four to forty-eight hours after completion of each conditioning regimen, patients will receive a transplant of a CD34+ progenitor cell-enriched, T-cell depleted fraction of GCSF-mobilized PBSC after fractionation on the CliniMACS device, from his/her HLA compatible donor. Due to stringent T-cell depletion, no significant Graft-versus-host disease is anticipated. Should Graft-versus-host disease occur, standard treatment would be initiated per the Transplant Service guidelines.

The purpose of this trial is to evaluate the potential of T-cell depleted Haploidentical Stem Cell Transplant fractionated by the CliniMACS system, when administered for disease targeted cytoreductive regimens, to secure consistent engraftment and hematopoietic reconstitution in HLA-compatible related or unrelated hosts, and to prevent or abrogate acute and chronic forms of Graft-versus-host disease. This study seeks to validate that these pre-transplant conditioning regimens, when administered with a CD34+ progenitor cell enriched, T-cell depleted graft, fractionated in the CliniMACS system, will be associated with a low incidence of non-leukemic mortality.

The sample size is as follows:

Regimen A: Hyperfractionated Total Body Irradiation/Thiotepa/Cyclophosphamide: 100 patients Regimen B: Busulfan/Melphalan/Fludarabine: 100 patients It is anticipated that the accrual will last five years. Patients will be followed for two years following transplantation.

ELIGIBILITY:
Inclusion Criteria:

Malignant conditions or other life-threatening disorders correctable by transplant for which CD34+ selected, T-cell depleted allogeneic hematopoietic stem cell transplantation is indicated such as:

1. Acute myeloid leukemia (AML) in 1st remission - for patients who is AML does not have 'good risk' cytogenetic features (i.e. t8:21, t 15: 17, inv16).
2. Secondary AML in 1st remission
3. AML in 1st relapse or 2nd remission
4. Acute lymphoblastic leukemia (ALL) / Chronic Lymphocytic Leukemia (CLL) in pt remission clinical or molecular features indicating a high risk for relapse; or ALL/CLL 2nd remission
5. Chronic myelogenous leukemia (CML) failing to respond to or not tolerating Imatinib or Dasatinib in first chronic phase of disease; CML in accelerated phase, second chronic phase, or in CR after accelerated phase or blast crisis.
6. Non-Hodgkin's lymphoma with chemo responsive disease in any of the following categories:

   1. Intermediate or high-grade lymphomas who have failed to achieve a first CR or have relapsed following a 1st remission who are not candidates for autologous transplants.
   2. Any NHL in remission which is considered not curable with chemotherapy alone and not eligible/appropriate for autologous transplant.
7. Myelodysplastic syndrome (MDS): RA/RARS/RCMA with high-risk cytogenetic features or transfusion dependence, as well as RAEB-1 and RAEB-2 and Acute Myelogenous Leukemia (AML) evolved from MDS.
8. Chronic myelomonocyte leukemia: CMML-1 and CMML-2.
9. Multiple Myeloma with disease in the following categories:

   1. Patients with relapsed multiple myeloma following autologous stem cell transplantation who have achieved at least partial response following additional chemotherapy.
   2. Patients with high-risk cytogenetics at diagnosis must have achieved at least a partial response following autologous stem cell transplantation. Patients must have complex karyotype, del l7p, t4; 14 and/or t 4; 16 by Fluorescence in situ hybridization (FISH) and/or del l3 by karyotyping.

The following inclusion criteria are also required:

* Patient's age includes from birth on to < 74 years old.
* Patients may be of either gender or any ethnic background.
* Patients must have a Karnofsky (adult) Performance Status of at least 70%
* Patients must have adequate organ function measured by:

Cardiac: asymptomatic or if symptomatic then LVEF at rest must be 50% and must improve with exercise.

Hepatic: < 3x ULN AST and: s 1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia or if the hyperbilirubinemia is directly caused by the disease in which the patient is receiving a transplant (e.g. AML Chloroma obstructing the biliary tree). Patients with higher bilirubin levels due to causes other than active liver disease is also eligible with Pl approval e.g. patients with PNH, Gilbert's disease or other hemolytic disorders.

Renal: serum creatinine: s; 1.2 mg/di or if serum creatinine is outside the normal range, then CrCl > 40 ml/m in (measured or calculated/estimated).

Pulmonary: asymptomatic or if symptomatic, DLCO 50% of predicted (corrected for hemoglobin).

Each patient must be willing to participate as a research subject and must sign an informed consent form.

Donor Inclusion Criteria

* Each donor must meet criteria outlined by institutional guidelines
* Donor should agree to undergo general anesthesia and bone marrow harvest collection if PBSC yield is inadequate or otherwise not transplantable for whatever reason.

Exclusion Criteria:

Subject Exclusion Criteria

* Female patients who are pregnant or breast-feeding
* Active viral, bacterial or fungal infection
* Patient seropositive for HI V-I /II; HTLV -I /II
* Presence of leukemia in the CNS.

Donor Exclusion Criteria

• If donors do not meet institutional guidelines, exclusion will be considered.

Max Age: 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Assess the change of incidence and severity of chronic GvHD | 6 months, 1 year, 2 years
  To assess the incidence and severity of chronic GvHD following T cell depleted, CD34+ progenitor cell enriched transplants fractionated by the CliniMACS system.
Assess the change of incidence and severity of acute GvHD | 6 months, 1 year, 2 years
  To assess the incidence and severity of acute GvHD following T cell depleted, CD34+ progenitor cell enriched transplants fractionated by the CliniMACS system.
Assess the change of incidence of non-relapse mortality | 6 months, 1 year, 2 years
  To assess the incidence of non-relapse mortality (transplant-related mortality) following each cytoreduction regimen and a transplant fractionated by the CliniMACS system.
Estimate the probability change of survival and disease-free survival (DFS) | 6 months, 1 year, 2 years
  To estimate the probability of survival and disease-free survival (DFS) at 6 months, 1 year and 2 years post-transplant for each disease-targeted cytoreduction regimen when used with a T-cell depleted graft fractionated by the CliniMACS system.

SECONDARY OUTCOMES:
Determine the proportion of patients receiving optimal CD34+; CD3+ | 6 months, 1 year, 2 years
  To determine the proportion of patients receiving optimal CD34+ (>5x 106/kg) and CD3+ (< 5 x104/kg) cell doses the proportion recurring suboptimal doses (<3 x 106/kg) CD34+ cells; and the proportion of patients receiving CD3+ T-cell doses >5 x 104/kg.
Correlate doses of CD34+ progenitors and CD3+ T cells with engraftment | 6 months, 1 year, 2 years
  To correlate doses of CD34+ progenitors and CD3+ T cells with engraftment, graft vs. host disease and non-relapse mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Koehne, MD, Principal Investigator — Miami Cancer Institute (MCI) at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute at Baptist Health, Inc., Miami, Florida, United States

REFERENCES:
- See also: MCI - Website — http://baptisthealth.net/cancer-care/home